CLINICAL TRIAL: NCT02542384
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Adaptive Design Study Evaluating the Analgesic Efficacy and Safety of Intravenous CR845 in Patients Undergoing Abdominal Surgery
Brief Title: A Study Evaluating the Overall Pain Relief and Safety of Intravenous (IV) CR845 in Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-CLIN3001
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Post Abdominal Surgery Pain
Keywords: abdominal surgery; laparoscopy; Hysterectomy; Prostatectomy; Hemi-colectomy; Ventral Hernia repair; CR845; analgesic; kappa opioid; partial bowel resection; difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CR845 IV 1 mcg/kg (Active Comparator): CR845 IV solution will be supplied in 2 mL glass vials.Study drug will be administered as an IV bolus into an infusion line, the volume is dependent upon the patient's body weight.
  Interventions: Drug: CR845 IV 1 mcg/kg
- CR845 IV 0.5 mcg/kg (Active Comparator): CR845 solution will be supplied in 2 mL glass vials. Study drug will be administered as an IV bolus into an infusion line, the volume is dependent upon the patient's body weight.
  Interventions: Drug: CR845 IV 0.5 mcg/kg
- Placebo IV (Placebo Comparator): Placebo will be supplied in matched vials containing the same volume of buffer but with no active drug. It will be administered as an IV bolus into an infusion line, the volume is dependent upon the patient's body weight.
  Interventions: Drug: Placebo IV

INTERVENTIONS:
Drug: CR845 IV 1 mcg/kg — CR845 IV 1 mcg/kg will be administered as an IV bolus 2x loading dose one hour prior to anesthetic induction for surgery, then a dose within 30 minutes of the patient being considered stable in the post operative recovery room. Subsequent dosing will be administered at 6, 12 and 18 hours.
  Antinausea rescue medication (ondansetron 4 mg IV) may be requested, as well as analgesic rescue medication (morphine 5mg IV), post surgery, as needed. Saline infusion (IV 0.45%) for fluid replenishment will be provided.
  Arms: CR845 IV 1 mcg/kg
Drug: CR845 IV 0.5 mcg/kg — CR845 IV 0.5 mcg/kg will be administered as an IV bolus 2x loading dose one hour prior to anesthetic induction for surgery, then a dose within 30 minutes of the patient being considered stable in the post operative recovery room. Subsequent dosing will be administered at 6, 12 and 18 hours.
  Antinausea rescue medication (ondansetron 4 mg IV) may be requested, as well as analgesic rescue medication (morphine 5mg IV), post surgery, as needed.
  Saline infusion (IV 0.45%) for fluid replenishment will be provided.
  Arms: CR845 IV 0.5 mcg/kg
Drug: Placebo IV — Placebo IV will be administered as an IV bolus 2x loading dose one hour prior to anesthetic induction for surgery, then a dose within 30 minutes of the patient being considered stable in the post operative recovery room. Subsequent dosing will be administered at 6, 12 and 18 hours.
  Antinausea rescue medication (ondansetron 4 mg IV) may be requested, as well as analgesic rescue medication (morphine 5mg IV), post surgery, as needed.
  Saline infusion (IV 0.45%) for fluid replenishment will be provided.
  Arms: Placebo IV

SUMMARY:
The study schedule is comprised of a 14-day Screening Period, a treatment period and an observation period. All eligible subjects will be randomized into one of 3 treatment groups (1 of 2 dose levels or matched placebo). Study drug CR845 will be administered intravenously prior to surgery, and at specific time intervals post surgery. Additional rescue pain and anti-nausea medication will be made available. Post surgical changes in pain intensity, nausea and vomiting will be assessed.

DETAILED DESCRIPTION:
Patients will be admitted to the surgical center on the day of their abdominal surgery (Day 1, unless admission the night before is required). All patients will be seen by the study staff to confirm eligibility, review study procedures, and conduct all pre-surgical assessments required for randomization.

Qualified patients will be randomized into 1 of 3 treatment groups, corresponding to 1 of 2 dose levels of intravenous (IV) CR845 (0.5 or 1 mcg/kg) or matched placebo, respectively.

Study drug will be administered every 6 hours during the 24-hour post-operative treatment period following these initial 2 drug administrations:

* Pre-Operative dose: Within one hour prior to anesthetic induction for surgery. This dose will be a 2X loading dose.
* Baseline post-operative dose: within 30-minutes of being considered stable in the Post-Anesthesia Care Unit (PACU)

Subsequent dosing will be administered at 6, 12 and 18 hours.

During the Treatment and Observation Period, pain intensity scores will be obtained at specified time points and episodes of nausea or vomiting will be recorded. Upon request, patients may be provided with analgesic or anti-nausea rescue medication (restricted to morphine (if tolerated), and ondansetron, respectively) at any time after the Baseline dose of study drug is administered.

Blood sampling and safety assessments will be conducted during this period as well.

Patients will remain in the hospital until Day 3 (48-hours after surgery) at which point they will be evaluated for discharge. A follow-up medical evaluation will be scheduled within 7 - 10 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

- A patient will be eligible for study participation if the subject meets the following criteria:

1. Voluntarily provide written informed consent to participate in the study prior to any study procedures.
2. Able to speak, read, and communicate clearly in English or Spanish; able to read and understand the study procedures.
3. Male or female between 21 and older at the time of Screening.
4. Scheduled for abdominal surgery (hysterectomy; prostatectomy; hemi-colectomy (including partial bowel resections) or ventral hernia repair) with no collateral procedures.
5. Patient is categorized as American Society of Anesthesiologists (ASA) risk class of I, II or III.
6. Has a body mass index (BMI) within 18.0-40.0 kg/m2 and weight between 50 kg and 112 kg, inclusive.
7. For women of childbearing potential- has a negative result on serum pregnancy testing at Screening and urine pregnancy test at Admission and does not currently breast feed, or is planning to do so within 30 days of receiving the last dose of study drug.
8. If female, the patient must be:

   * Of childbearing potential and practicing an acceptable form of birth control (defined as the use of an intrauterine device; a barrier method with spermicide; condoms, any form of hormonal contraceptives; or abstinence from sexual intercourse) for 3 days following the last dose of study drug.
   * Of non-childbearing potential defined as surgically or biologically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or postmenopausal for at least 1 year).
9. If male, the patient must be surgically or biologically sterile. If not sterile, the patient must agree to use an acceptable form of birth control with heterosexual partner (as described in inclusion criteria #8a) or abstain from sexual relations for 3 days following the last dose of study drug.
10. Is free of other physical, mental, or medical conditions, which, in the opinion of the Investigator, would make study participation inadvisable.
11. Following surgery, the patient will be eligible for the second dose of study drug.

Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

1. Has a serum sodium level > 143 mmol/L at Screening.
2. Has a serum sodium level < 136 mmol/L at Screening.
3. Patient is unwilling or unable to comply with the study procedures and assessments until the end of the 48-hour treatment and observation period.
4. Has moderate to severe obstructive sleep apnea, which, in the opinion of the Investigator is not being adequately treated (i.e., Nasal/Facial C-PAP), and will pose an unacceptable risk.
5. Has known allergies or hypersensitivity to drugs that may be used during the study, including those used during the surgical procedure and in the post-operative period [e.g., inhaled anesthetics (such as sevoflurane), midazolam, opioids (such as fentanyl and morphine sulfate), propofol or other sedatives, local anesthetics, antiemetics (such as ondansetron) non- steroidal anti-inflammatory drugs (such as ketorolac) or acetaminophen].
6. Uses antipsychotics, antiepileptics, sedatives, hypnotics, or antianxiety agents, selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants with a dose change < 30 days prior to surgery.
7. Has a history or current diagnosis of substance dependence (except caffeine or nicotine) or alcohol abuse, according to the criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
8. Has a positive urine drug screen for drugs of abuse at Screening.
9. Is unwilling to abstain from alcohol consumption for a period beginning 24 hours prior to Admission until the time of Discharge from the hospital.
10. Suffers from chronic dizziness, vestibular disorders, or has experienced severe continuous diarrhea, retching, vomiting, or moderate or severe nausea and/or dizziness for any reason within 72 hours prior to Admission.
11. Has been diagnosed with a condition of hyperhidrosis (excessive sweating) or primary hypodipsia (abnormally diminished thirst).
12. Has donated or had significant loss of whole blood (240 mL or more) within 30 days or plasma within 14 days prior to Admission.
13. Has a history (within 6 months) of clinically meaningful orthostatic changes in vital signs - OR - a decrease in systolic blood pressure by > 20 mm Hg or a decrease in diastolic blood pressure by 10 mm Hg together with an increase in heart rate of > 30 beats per minute when transitioning from supine to standing measurements at the time of Screening.
14. Hasmedicalconditions(e.g.,cardiovascular,pulmonary,hepatic,renal, hematologic, gastrointestinal, endocrine (adrenal hyperplasia), immunologic, dermatologic, neurologic, oncologic or psychiatric condition) or a significant laboratory abnormality that, in the Investigator's opinion, would jeopardize the safety of the patient or is likely to confound the study measurements.
15. Has congestive heart failure.
16. Has taken any diuretic medications within 2-weeks prior to the scheduled surgery.
17. Has an oxygen saturation < 92% on room air at Screening or Admission.
18. Has impaired renal function indicated by serum creatinine greater than 2 times the reference upper limit of normal (ULN).
19. Has a serum alanine aminotransferase (ALT) or aspartate aminotransferase AST) greater than 2.5 times the reference upper limit of normal (ULN), or total bilirubin greater than 2 times the ULN at Screening.
20. Has, in the opinion of the Investigator, any clinical signs of dehydration or hypovolemia (e.g., symptomatic hypotension) or associated laboratory abnormalities, e.g., elevated hematocrit, elevated blood urea nitrogen (BUN) >1.5 x the reference ULN at Screening.
21. Has taken opioid analgesics for more than 10 consecutive days for any reason within the past 3 months prior to Screening.
22. Has taken opioid or non-opioid pain medication (e.g., NSAIDs such as naproxen, cyclooxygenase-2 inhibitors) within the 12 hours prior to surgery.
23. Has received another investigational drug within 30 days prior to Admission or has planned to participate in another clinical trial while enrolled in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
A comparison of the change in Pain Intensity over time using the Numeric Rating Scale | 24 hours
  Using the Numeric Rating Scale (NRS) to quantify the difference between CR845-treated patients and placebo-treated patients.

SECONDARY OUTCOMES:
A study of the comparison of Post Surgical Nausea and Vomiting (PONV) scores | 6 hours
  Incidence of vomiting will be analyzed against placebo
A comparison of the number of rescue medication doses administered | 24 hours
  Count the number of rescue medication doses administered following surgery for the CR845 IV patients vs Placebo-treated patients
Patient Global Assessment of study drug | 24 hours (or early termination)
  Patients will complete a PGA (Patient Global Assessment) of the study drug.

OTHER OUTCOMES:
Ongoing safety evaluation of CR845 assessed by physical examination, adverse events, vital signs, and laboratory evaluations | 10 Days
  The safety of CR845 in this patient population will be assessed by physical examination, monitoring of adverse events, vital signs, fluid balance, and laboratory evaluations at specified times. Participants with clinically significant lab values or abnormal exam findings, as well as those with adverse events found to be related to the study drug will be compared to those receiving placebo.
  Safety data will be reviewed on an ongoing basis by the sponsor and an Independent Data Monitoring Committee (IDMC).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Stauffer, DO, MBA, Study Director — Cara Therapeutics
Locations (23):
- United States (23):
  - Cara Therapeutics Study Site, Sheffield, Alabama
  - Cara Therapeutics Study Site, New Haven, Connecticut
  - Cara Therapeutics Study Site, Bradenton, Florida
  - Cara Therapeutics Study Site, Gainesville, Florida
  - Cara Therapeutics Study Site, Maitland, Florida
  - Cara Therapeutics Study Site, Miami Gardens, Florida
  - Cara Therapeutics Study Site, Pensacola, Florida
  - Cara Therapeutics Study Site, St. Petersburg, Florida
  - Cara Therapeutics Study Site, Chicago, Illinois
  - Cara Therapeutics Study Site, Boston, Massachusetts
  - Cara Therapeutics Study Site, Camden, New Jersey
  - Cara Therapeutics Study Site, Neptune City, New Jersey
  - Cara Therapeutics Study Site, Durham, North Carolina
  - Cara Therapeutics Study Site, Cleveland, Ohio
  - Cara Therapeutics Study Site, Columbus, Ohio
  - Cara Therapeutics Study Site, Pittsburgh, Pennsylvania
  - Cara Therapeutics Study Site, Chattanooga, Tennessee
  - Cara Therapeutics Study Site, Bellaire, Texas
  - Cara Therapeutics Study Site, Fort Worth, Texas
  - Cara Therapeutics Study Site, Houston, Texas
  - Cara Therapeutics Study Site, Plano, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Salt Lake City, Utah